CLINICAL TRIAL: NCT02628782
Title: InSeal VCD Large Bore Vascular Closure Device Clinical Study
Brief Title: InSeal VCD Large Bore Vascular Closure Device Safety and Effectiveness Clinical Study
Acronym: InSealVCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSeal Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-14-003I
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2019-01

CONDITIONS: Percutaneous Closure of Artery Access Sites
Keywords: large bore endovascular catheterization procedures; Vascular Closure Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- InSeal VCD (Experimental): InSeal's Vascular Closure Device Use of the experimental VCD to close the access site of the artery
  Interventions: Device: InSeal's Vascular Closure Device

INTERVENTIONS:
Device: InSeal's Vascular Closure Device — Intravascular closure device

SUMMARY:
The InSeal vascular closure device (VCD) is assessed as percutaneous closure of artery access sites for quick hemostasis and ambulation in patients who have undergone large bore endovascular catheterization procedures.

The study hypothesis is that the VCD is safe and efficient in achieving hemostasis in the study population.

DETAILED DESCRIPTION:
The increasing variety of arterial devices having a large crossing profile requiring the use of a large bore sheath is mandating focus on large bore closure. Such procedures include endovascular abdominal repair (EVAR), thoracic (TEVAR) aortic repairs and transcatheter aortic valve implantation (TAVI) typically involve sheaths and delivery catheters with 14-25Fr profiles.

Today, the typical closing technique (labeled in Europe) for such large sheath size is a one where sutures are deployed prior to the insertion of the large sheath with the sutures tied at the end of the procedure. This technique is cumbersome, hard to learn, complex to use and has relative high complications and failure rate.

The InSeal VCD device model 13-517, is easy to use, fast, affords immediate reliable hemostasis, and supports a wide range of sheath punctures size and artery's dia. 6-10 mm, while leaving a minimal amount material behind and will not limit re-access.

While each of these features may be found in one commercial device or another, to date there is no single device that meets all the market requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for large bore catheterization procedure (such as TAVI, aortic endograft repair) using a CE approved 18Fr access sheath.
2. Femoral, axillary or subclavian artery diameter at sheath insertion site is between 5.5-10mm
3. Subject age is at least 18 years
4. Patient has signed most recent approved version of the Informed Consent
5. Existence of an additional arterial access port is required in instances where an occluding balloon is planned to be used as a safety precaution.

Exclusion Criteria:

1. Women Of Child Bearing Potential (WOCBP)
2. Legally non-competent patients
3. Patient participating in another clinical study at the time of the InSeal VCD study
4. Sheath insertion point is less than 12mm proximal to a bifurcation having a diameter greater than 2.5mm
5. Side branch of greater than 2.5mm in diameter less than 4cm proximal to the puncture site.
6. Known severe allergy to metal and membrane material
7. Prior target artery closure with a vascular closure device having intravascular component (such as Angio-Seal) 30 days prior to catheterization
8. Subjects with known coagulopathy, preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the vessel access site prior to artery closure
9. Patients that do not tolerate aspirin and clopidogrel anticoagulation treatment
10. Prior vascular surgery or vascular graft in region of access site
11. Significant calcification, atherosclerotic disease, or stent within 1.5 cm of the puncture site that may interfere with the operation of the experimental device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Hemostasis within 15 minutes | 15 minutes
  Hemostasis within 15 minutes following vessel access site closure and after ACT falls below 200 seconds. Measured by operator using standard time measuring device (e.g., stopwatch)

SECONDARY OUTCOMES:
Combined rate of closure-device related major adverse events | 1 month
  Combined rate of closure-device related major adverse events in first month as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ran Kornowski, MD, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky